CLINICAL TRIAL: NCT02559596
Title: Reactivation of Varicella Zoster Virus and Risk of Vascular Disease in the Health Survey for England: a Nested Case Control Study
Brief Title: Reactivation of Varicella Zoster Virus and Risk of Vascular Disease
Status: Withdrawn | Type: Observational
Why Stopped: Linked data not available for research within requisite time period
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 15/0311; F192 (Other Grant/Funding Number: University College London Hospitals BRC)
Record Dates: First submitted 2015-09-23; First posted 2015-09-24 (Estimated); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Varicella Zoster; Stroke; Transient Ischaemic Attack; Acute Myocardial Infarction
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases: Adults (aged 16+) with stored serum samples collected for the Health Survey for England (HSE) between 2009 and 2013, who have a record of hospitalisation for stroke, transient ischaemic attack or myocardial infarction occurring after their participation in the HSE.
- Controls: Adults (aged 16+) with stored serum samples collected for the Health Survey for England (HSE) between 2009 and 2013, who do not have a record of hospitalisation for stroke, transient ischaemic attack or myocardial infarction and are matched to cases on age, gender and year of participation in the HSE.

SUMMARY:
The purpose of this study is to investigate whether there is an association between stroke or heart attack and reactivation of varicella zoster virus, measured by antibody levels, using linked data from the Health Survey for England and secondary care.

DETAILED DESCRIPTION:
This study will use a case control design to investigate whether adult participants in the Health Survey for England between 2009 and 2013 who were admitted to hospital with either a stroke or heart attack had higher preceding levels of varicella zoster virus antibodies measured in stored serum samples compared to matched controls with no history of heart attack or stroke, controlling for a range of potential demographic, lifestyle and clinical confounders.

This study is funded by the University College London Hospitals Biomedical Research Centre Fast Track grant scheme and has received ethics approval (ref 15/NW/0456).

ELIGIBILITY:
Inclusion Criteria:

* Previous participant in the HSE between 2009 and 2013 with stored serum available.
* Either a record of stroke or TIA or MI in linked HES data between 01/01/2009 and 31/12/2013 or selected as a matched control for those with a record of stroke/ TIA/MI in HES data.
* Male or female, aged 16 years or above.

Exclusion Criteria:

* HSE participant with no stored serum sample

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be drawn from adults who have already participated in the Health Survey for England between 2009 and 2013 and who have a stored serum sample available for analysis. No new participants will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Odds ratio for the effect of high serum antibody titre on stroke or other vascular outcomes | Outcome assessed within 5 years of serum sample

SECONDARY OUTCOMES:
Prevalence of age- and sex-specific serum VZV antibody titres as a marker for virus reactivation | Assessed at baseline recruitment to the HSE

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Warren-Gash, MRCP PhD, Principal Investigator — UCL